CLINICAL TRIAL: NCT01132118
Title: Hydroxychloroquine to Improve Insulin Sensitivity in Rheumatoid Arthritis
Acronym: RA PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Director of Clinical Sciences, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P001926; R21AR057924 (NIH)
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis; Insulin Resistance
Keywords: rheumatoid arthritis; insulin resistance; hydroxychloroquine; cholesterol
MeSH Terms: conditions — Arthritis, Rheumatoid; Insulin Resistance | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo then HCQ (Other): This arm of the study will contain half the study population after randomization. The participants in this arm will receive hydroxychloroquine for 8 weeks and then crossover to a placebo for 8 weeks. Study staff will be blinded to which order they are taking the hydroxychloroquine and placebo in.
  Interventions: Drug: Hydroxychloroquine
- HCQ then Placebo (Other): This arm of the study will contain half the study population after randomization. The participants in this arm will receive hydroxychloroquine for 8 weeks and then crossover to a placebo for 8 weeks. Study staff will be blinded to which order they are taking the hydroxychloroquine and placebo in.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine comes in 200 mg tablets and is taken orally. The dose provided will be based upon a calculation of 6.5 mg/kg (subject's weight), which is the dose range commonly used to treat rheumatoid arthritis and lupus. Dosages will be rounded to the nearest 100 mg.
  Other Names: Plaquenil

SUMMARY:
The purpose of this study is to determine whether hydroxychloroquine (HCQ) reduces insulin resistance in non-diabetic subjects with rheumatoid arthritis (RA). The investigators will conduct a double-blind randomized crossover trial in subjects with RA to test the hypothesis that HCQ improves insulin sensitivity. The investigators will also use data from the trial to identify determinants of insulin resistance in RA. The investigators hypothesize that RA will be associated with an increased risk of insulin resistance and that independent risk factors for increased insulin resistance in RA include higher BMI, elevated acute phase reactants, greater fat to muscle ratio, and less physical activity.

DETAILED DESCRIPTION:
Our ability to better control the pain and disability of rheumatoid arthritis (RA) now focuses attention on reducing the impact of RA-associated comorbidities. The most common cause of death in RA is cardiovascular (CV) disease, and the risk of myocardial infarction and stroke are approximately doubled in RA. The determinants of CV risk in RA include traditional CV risk factors as well as aspects of the inflammatory process defining RA. It is likely that RA-associated inflammation accelerates atherosclerosis through direct effects on the endothelium as well as indirect effects on insulin metabolism. Several studies report an increased prevalence of insulin resistance among persons with RA. However, it is not clear whether the inflammation of RA causes insulin resistance. Corticosteroids and abnormalities in the hypothalamic-pituitary axis may also contribute to abnormal glucose metabolism. Little information is available to guide management of a pre-diabetic insulin resistance state in RA.

Hydroxychloroquine (HCQ), a commonly used medicine early in RA, may play a role in improving insulin resistance. Several previous trials demonstrated the ability of HCQ to reduce blood glucose levels in diabetics, and a large epidemiologic study found that subjects with RA using HCQ were less likely to develop diabetes. In animal models, anti-malarials lower blood glucose through slowing insulin metabolism.

With CV disease a major comorbidity in RA and insulin resistance possibly a major determinant of CV risk, intervention studies need to begin to translate prior work into clinical therapeutics.

Relevance: If this study demonstrates a beneficial effect of HCQ on insulin resistance among the randomized subjects, this would provide strong evidence that HCQ has benefits beyond RA and SLE disease activity. Currently, HCQ is stopped in many patients as they "step-up" to more aggressive DMARD treatments, or HCQ may never be tried in some patients who present with RA carrying with poor prognosis. If HCQ improves insulin sensitivity, there may be rationale for continuing HCQ chronically in patients with RA. As well, a larger clinical endpoint study would be strongly considered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide informed consent and comply with study visits
* Hemoglobin ≥ 10 g/dL (within last two months)
* WBC ≥ 4 K/uL (within last two months)
* Platelet count ≥ 150 ≤ 450 K/uL (within last two months)
* (GFR) Creatinine clearance ≥ 70 ml/min (MDRD) (within last two months)
* SGOT, SGPT ≤ 1.5 times upper limits of normal (within last two months)
* Normal eye exam within 12 months of study entry (copy of letter from subject's ophthalmologist or optometrist stating that the subject has no evidence of macular pathology)
* Diagnosis of rheumatoid arthritis

Exclusion Criteria:

* History of any neuromuscular disease including muscular dystrophy, metabolic myopathies, peripheral neuropathy, multiple sclerosis, and other myopathies or myositides
* History of diabetes or fasting plasma glucose of 126 mg/dl or greater
* History of any untoward reaction to antimalarials
* Uncontrolled hypertension (>140/90)
* History of any ophthalmologic disease except for glaucoma or cataracts
* Planned elective surgery during the study period
* Digoxin therapy
* Treatment with corticosteroids (> 5 mg) for any disorder
* History of psoriasis
* Any chronic disease that in the opinion of the investigator warrants exclusion (e.g. inflammatory bowel disease, malignancy other than basal cell carcinoma, chronic liver disease)
* History of chronic intestinal disorders (Crohn's disease, ulcerative colitis, celiac sprue, collagenous colitis, eosinophilic enteritis)
* Creatinine clearance ≤ 60 ml/min (MDRD) (within last two months)
* Hemoglobin ≤ 10 g/dL (within last two months)
* WBC ≤ 4 K/uL (within last two months)
* Platelet count ≤ 150 ≥ 450 K/uL (within last two months)
* SGOT, SGPT ≥ 1.5 times upper limits of normal (within last two months)
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Solomon, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Elena M Massarotti, MD, Principal Investigator — Brigham and Women's Hospital; Rajesh K Garg, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] Reilly MP, Wolfe ML, Rhodes T, Girman C, Mehta N, Rader DJ. Measures of insulin resistance add incremental value to the clinical diagnosis of metabolic syndrome in association with coronary atherosclerosis. Circulation. 2004 Aug 17;110(7):803-9. doi: 10.1161/01.CIR.0000138740.84883.9C. Epub 2004 Aug 2. PMID 15289378
- [Background] Hanley AJ, Williams K, Stern MP, Haffner SM. Homeostasis model assessment of insulin resistance in relation to the incidence of cardiovascular disease: the San Antonio Heart Study. Diabetes Care. 2002 Jul;25(7):1177-84. doi: 10.2337/diacare.25.7.1177. PMID 12087016
- [Background] Glaser K, Sung ML, O'Neill K, Belfast M, Hartman D, Carlson R, Kreft A, Kubrak D, Hsiao CL, Weichman B. Etodolac selectively inhibits human prostaglandin G/H synthase 2 (PGHS-2) versus human PGHS-1. Eur J Pharmacol. 1995 Jul 25;281(1):107-11. doi: 10.1016/0014-2999(95)00302-2. PMID 8566109
- [Background] Gabriel SE. The epidemiology of rheumatoid arthritis. Rheum Dis Clin North Am. 2001 May;27(2):269-81. doi: 10.1016/s0889-857x(05)70201-5. PMID 11396092
- [Background] Young A, Koduri G, Batley M, Kulinskaya E, Gough A, Norton S, Dixey J; Early Rheumatoid Arthritis Study (ERAS) group. Mortality in rheumatoid arthritis. Increased in the early course of disease, in ischaemic heart disease and in pulmonary fibrosis. Rheumatology (Oxford). 2007 Feb;46(2):350-7. doi: 10.1093/rheumatology/kel253. Epub 2006 Aug 14. PMID 16908509
- [Background] Goodson N, Marks J, Lunt M, Symmons D. Cardiovascular admissions and mortality in an inception cohort of patients with rheumatoid arthritis with onset in the 1980s and 1990s. Ann Rheum Dis. 2005 Nov;64(11):1595-601. doi: 10.1136/ard.2004.034777. Epub 2005 Apr 20. PMID 15843450
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Maradit-Kremers H, Nicola PJ, Crowson CS, Ballman KV, Gabriel SE. Cardiovascular death in rheumatoid arthritis: a population-based study. Arthritis Rheum. 2005 Mar;52(3):722-32. doi: 10.1002/art.20878. PMID 15751097
- [Background] Solomon DH, Curhan GC, Rimm EB, Cannuscio CC, Karlson EW. Cardiovascular risk factors in women with and without rheumatoid arthritis. Arthritis Rheum. 2004 Nov;50(11):3444-9. doi: 10.1002/art.20636. PMID 15529391
- [Background] Ridker PM, Stampfer MJ, Rifai N. Novel risk factors for systemic atherosclerosis: a comparison of C-reactive protein, fibrinogen, homocysteine, lipoprotein(a), and standard cholesterol screening as predictors of peripheral arterial disease. JAMA. 2001 May 16;285(19):2481-5. doi: 10.1001/jama.285.19.2481. PMID 11368701
- [Background] Dessein PH, Joffe BI. Insulin resistance and impaired beta cell function in rheumatoid arthritis. Arthritis Rheum. 2006 Sep;54(9):2765-75. doi: 10.1002/art.22053. PMID 16947779
- [Background] Chung CP, Oeser A, Solus JF, Gebretsadik T, Shintani A, Avalos I, Sokka T, Raggi P, Pincus T, Stein CM. Inflammation-associated insulin resistance: differential effects in rheumatoid arthritis and systemic lupus erythematosus define potential mechanisms. Arthritis Rheum. 2008 Jul;58(7):2105-12. doi: 10.1002/art.23600. PMID 18576352
- [Background] Quatraro A, Consoli G, Ceriello A, Giugliano D. Is there a role for chloroquine treatment in diabetes? A three case report. Diabete Metab. 1988 Sep-Oct;14(5):666-7. No abstract available. PMID 3069509
- [Background] Garcia-Webb P, Bonser AM. Insulin binding and degradation in isolated hepatocytes from streptozotocin injected rats. Biochem Biophys Res Commun. 1985 Apr 30;128(2):487-93. doi: 10.1016/0006-291x(85)90073-7. PMID 3888217
- [Background] Emami J, Pasutto FM, Mercer JR, Jamali F. Inhibition of insulin metabolism by hydroxychloroquine and its enantiomers in cytosolic fraction of liver homogenates from healthy and diabetic rats. Life Sci. 1999;64(5):325-35. doi: 10.1016/s0024-3205(98)00568-2. PMID 10072192
- [Background] Quatraro A, Consoli G, Magno M, Caretta F, Nardozza A, Ceriello A, Giugliano D. Hydroxychloroquine in decompensated, treatment-refractory noninsulin-dependent diabetes mellitus. A new job for an old drug? Ann Intern Med. 1990 May 1;112(9):678-81. doi: 10.7326/0003-4819-112-9-678. PMID 2110430
- [Background] Gerstein HC, Thorpe KE, Taylor DW, Haynes RB. The effectiveness of hydroxychloroquine in patients with type 2 diabetes mellitus who are refractory to sulfonylureas--a randomized trial. Diabetes Res Clin Pract. 2002 Mar;55(3):209-19. doi: 10.1016/s0168-8227(01)00325-4. PMID 11850097
- [Background] Wasko MC, Hubert HB, Lingala VB, Elliott JR, Luggen ME, Fries JF, Ward MM. Hydroxychloroquine and risk of diabetes in patients with rheumatoid arthritis. JAMA. 2007 Jul 11;298(2):187-93. doi: 10.1001/jama.298.2.187. PMID 17622600
- [Derived] Solomon DH, Garg R, Lu B, Todd DJ, Mercer E, Norton T, Massarotti E. Effect of hydroxychloroquine on insulin sensitivity and lipid parameters in rheumatoid arthritis patients without diabetes mellitus: a randomized, blinded crossover trial. Arthritis Care Res (Hoboken). 2014 Aug;66(8):1246-51. doi: 10.1002/acr.22285. PMID 24470436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 potentially eligible RA patients were screened during 2010-2011. 7 subjects did not meet inclusion/exclusion criteria at screening and 63 declined participation.
Pre-assignment Details: 37 subjects were initially consented, 7 withdrew consent before randomization. Thirty patients were randomized. Five patients withdrew consent after randomization and two patients stopped participation in the study due to non-serious adverse events.
Groups:
- HCQ Then Placebo; Placebo Then HCQ: This arm of the study contains half the study population after randomization. The participants in this arm received hydroxychloroquine for 8 weeks and then crossed over to a placebo for 8 weeks. Study staff was blinded to which order they were taking the hydroxychloroquine and placebo in.
  Hydroxychloroquine: Hydroxychloroquine comes in 200 mg tablets and is taken orally. The dose provided will be based upon a calculation of 6.5 mg/kg (subject's weight), which is the dose range commonly used to treat rheumatoid arthritis and lupus. Dosages will be rounded to the nearest 100 mg.
Period: First Intervention (8 Weeks)
Arm/Group | HCQ Then Placebo | Placebo Then HCQ
Started | 15 | 15
Completed | 12 | 12
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Period: Second Intervention (8 Weeks)
Arm/Group | HCQ Then Placebo | Placebo Then HCQ
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were randomized to receive either HCQ or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | HCQ Then Placebo | Placebo Then HCQ | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 57 (14) | 56.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Index
Description: We will examine the effect of HCQ on the Matsuda Insulin Sensitivity Index (ISI) during the active treatment phase compared with placebo phase.
  ISI is based on insulin and glucose levels in a fasting state during an oral glucose tolerance test (OGTT) and is calculated as follows:
  ISI (Matsuda) = 10000/√ G0 X I0 X Gmean X Imean
  G0 - fasting plasma glucose (mg/dL) I0 - fasting plasma insulin (mIU/L) Gmean - mean plasma glucose during OGTT (mg/dL) Imean - mean plasma insulin during OGTT (mIU/L)
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: (dL x L)/(mg x mIU)
Groups:
- Hydroxychloroquine: This group contains results for when study participants were taking hydroxychlorquine.
  Hydroxychloroquine: Hydroxychloroquine comes in 200 mg tablets and is taken orally. The dose provided was based upon a calculation of 6.5 mg/kg (subject's weight), which is the dose range commonly used to treat rheumatoid arthritis and lupus. Dosages will be rounded to the nearest 100 mg.
- Placebo: This arm group contains the results for patients while they were on placebo.
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
(dL x L)/(mg x mIU)
  Baseline | 7.7 (4.8) | 7.7 (4.8)
  Period Value | 8.1 (4.5) | 7.8 (4.0)
  Change | 0.4 (2.9) | 0.14 (3.1)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; The P-value calculated was for the difference betweeen the change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.930, Wilcoxon (Mann-Whitney) — Unadjusted
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; The P-value was calculated for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.785, Regression, Linear — Adjusted for weight change

2. Secondary Outcome: HOMA-IR
Description: We will examine the effect of HCQ on HOMA-IR during the active treatment phase compared with placebo phase.
  HOMA-IR = (Glucose x insulin)/405
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: (mg x mIU)/(dL*L)
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
(mg x mIU)/(dL*L)
  Baseline | 2.0 (1.7) | 2.0 (1.7)
  Period | 1.7 (1.0) | 1.6 (0.79)
  Change | -0.3 (1.5) | -0.42 (1.4)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.575, Wilcoxon (Mann-Whitney) — Unadjusted P-value
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.308, Regression, Linear — Adjusted for weight change

3. Secondary Outcome: HOMA-B
Description: HOMA-B = (360 x Insulin)/(Glucose - 63)
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: (mIU x dL)/(L x mg)
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
(mIU x dL)/(L x mg)
  Baseline | 116.5 (100.4) | 116.5 (100.4)
  Period | 110.8 (81.6) | 109.7 (82.6)
  Change | -5.8 (72.9) | -6.8 (78.0)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference betweeen change during hydroxychloroquine versus placebo suing Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.468, Wilcoxon (Mann-Whitney) — Unadjusted
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.902, Regression, Linear — Adjusted for weight change

4. Secondary Outcome: Total Cholesterol
Description: mg/dL
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Baseline | 192.4 (37.5) | 192.4 (37.5)
  Period | 179.7 (44.3) | 189.4 (37.9)
  Change | -12.7 (20.0) | -3.0 (22.4)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney) — Unadjusted
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.004, Regression, Linear — Adjusted for weight change

5. Secondary Outcome: LDL Cholesterol
Description: mg/dL
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Baseline | 114.1 (29.8) | 114.1 (29.8)
  Period | 101.7 (36.7) | 109.9 (33.1)
  Change | -12.4 (20.1) | -4.2 (17.7)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney) — Unadjusted
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.011, Regression, Linear — Adjusted for weight change

6. Secondary Outcome: HDL Cholesterol
Description: mg/dL
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Baseline | 58.1 (17.9) | 58.1 (17.9)
  Period | 59.4 (18.2) | 60.3 (17.8)
  Change | 1.3 (6.7) | 2.2 (9.8)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.730, Wilcoxon (Mann-Whitney) — Unadjusted
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.208, Regression, Linear — Adjusted for weight change

7. Secondary Outcome: Triglycerides
Description: mg/dL
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Baseline | 100.6 (44.0) | 100.6 (44.0)
  Period | 92.4 (41.7) | 95.6 (44.9)
  Change | -8.2 (45.0) | -5.0 (20.1)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxychloroquine versus placebo using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.487, Wilcoxon (Mann-Whitney) — Unadjusted P-value
Statistical Analysis 2: Comparison: Hydroxychloroquine vs Placebo; P-value for the difference between the change during hydroxycholorquine versus placebo from a linear regression model; Test type: Superiority or Other; p = 0.884, Regression, Linear — P-value adjusted for weight change

ADVERSE EVENTS:
Groups:
- Hydroxychloroquine: Participants received hydroxychloroquine (HCQ) for 8 weeks.
  Hydroxychloroquine: Hydroxychloroquine comes in 200 mg tablets and is taken orally. The dose provided will be based upon a calculation of 6.5 mg/kg (subject's weight), which is the dose range commonly used to treat rheumatoid arthritis and lupus. Dosages will be rounded to the nearest 100 mg.
- Placebo: Participants received Placebo tablets for 8 weeks.
Arm/Group | Hydroxychloroquine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=15) | Placebo (N=15)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — 1 participants developed a rash when taking HCQ.
Liver Function Test Abnormality (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — 1 patient had abnormal liver function test scores while taking HCQ.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No